CLINICAL TRIAL: NCT06260501
Title: The Relationship Between Postoperative Complications and Wetting Solution-ideal Body Weight Ratio in Liposuction Procedures
Brief Title: Wetting Solution-ideal Body Weight Ratio in Liposuction Procedures
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Other Study IDs: ATADEK-2023-13/463
Record Dates: First submitted 2024-02-05; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Liposuction; Obesity; Postoperative Complications
Keywords: Liposuction; Obesity; Ideal body weight; Wetting solution; Epinephrine; Lidocaine
MeSH Terms: conditions — Obesity; Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High volume liposuction under general anesthesia with super-wet technique: Patients who underwent high-volume liposuction with super-wet technique using wetting-solution containing 0.5 gr lidocaine and 0.5 mg epinephrine in each liter under general anesthesia
  Interventions: Other: super-wet technique

INTERVENTIONS:
Other: super-wet technique — Liposuction with super-wet technique using wetting-solution containing 0.5 gr lidocaine and 0.5 mg epinephrine in each liter

SUMMARY:
Although the use of wetting solutions during high-volume liposuction is a standard approach, it is unclear how to optimize wetting solutions and components and their effect on postoperative complications.. Since the super-wet technique (aspiration of 1 cc per 1 cc of infiltrate) was introduced in 1986, it has become one of the most frequently applied techniques worldwide . Adrenaline and lidocaine are often added to WS due to their hemostatic and analgesic effects One of the major advantages of super-wet technique is that blood loss is quite low. However, potential cardiovascular side effects of WS and the amounts of epinephrine and lidocaine they contain, such as volume overload, local anesthetic toxicity, hypertension, arrhythmia, and tachycardia, are still a scoop of investigation. In this study, we examined the WS and the medications it contains from a different perspective to understand the possible cause of these adverse outcomes. Despite the most suitable candidates for liposuction are patients with a BMI<30 kg/m2 and low comorbidity and age, the patient group undergoing liposuction is often obese, and overweight individuals require that obesity-related pathophysiological changes be taken into consideration. Therefore, we analyzed the patients by dividing them into two groups according to the amount of WS applied according to their IBW (WS/IBW≤90ml/kg: group I and WS/IBW>90ml/kg: group I). In this study we aimed to evaluate the effect of wetting solutions and components calculated according to ideal body weight (IBW) on postoperative complications

DETAILED DESCRIPTION:
Liposuction is one of the most popular aesthetic surgical procedures worldwide making it possible to remove a significant amount of adipose tissue. Generally, liposuction is seen as a benign minor operation, but it can be considered a major surgery due to risk factors such as long operation times, intraoperative volume shifts, hypothermia, usage of high-dose adrenaline and lidocaine in wetting solution (WS), and possibly cardiac or pulmonary fatal complications. Therefore, anesthesiologists and plastic surgeons need to be aware of the intraoperative and postoperative pathophysiological changes caused by liposuction. In the literature, large-volume liposuction is defined as the removal of more than 5 liters of lipoaspirate in a single procedure.

The most suitable candidates for liposuction are individuals with BMI<30 kg/m2, but large-volume liposuction is applied more frequently to overweight and obese individuals. However, obesity can cause pathophysiological changes. In particular, increased cardiac output and changes in distribution volume may affect the pharmacokinetics and pharmacodynamics of drugs. Medications administered according to actual body weight (ABW) may lead to adverse outcomes due to overdose. For this reason, some approaches recommend adjusting perioperative medications according to IBW instead of ABW. The effects of WS and its components used in liposuction on patient outcomes have been examined in many studies, but the IBWs of the patients have not been taken into consideration. This study aimed to examine the effect of WSs calculated according to the IBW on postoperative complications and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society Of Anesthesiology physical status 1-3
* Patients who underwent high-volume liposuction with super-wet technique

Exclusion Criteria:

* Patients under 18 years of age
* Patients with a history of allergy to local anesthetic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent high-volume liposuction with super-wet technique under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Mean arterial pressure (MAP) was measured to detect hypertension and hypotension. | Duration of measurement was defined as one minute before anesthesia induction, during the surgery, and up to 2 days after surgery.
  MAP is a parameter used to evaluate blood pressure. If the MAP value was above 90 mm/hg, it was considered hypertension. If the MAP value was above 60 mm/hg, it was considered hypotension
The Numerical Pain Rating Scale (NRS) was used to assess postoperative pain level | Duration of measurement was defined as the period immediately after surgery and up to 2 days after the end of surgery.
  The Numerical Pain Rating Scale measures pain levels using a numerical scale from 0 to 10. 10 indicates the maximum value, and 0 indicates the minimum value. Values above 4 indicate a worse outcome, and values below 4 indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Serap Aktas Yildirim, M.D., Principal Investigator — Acibadem Mehmet Ali Aydinlar University School of Medicine, Department of Anesthesiology
Locations (1):
- Acibadem Altunizade Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Obara S, Yoshida K, Inoue S. How obesity affects the disposition of intravenous anesthetics. Curr Opin Anaesthesiol. 2023 Aug 1;36(4):414-421. doi: 10.1097/ACO.0000000000001280. Epub 2023 Jun 8. PMID 37314170
- [Background] Brown SA, Lipschitz AH, Kenkel JM, Sorokin E, Shepherd G, Grebe S, Oliver LK, Luby M, Rohrich RJ. Pharmacokinetics and safety of epinephrine use in liposuction. Plast Reconstr Surg. 2004 Sep 1;114(3):756-63; discussion 764-5. doi: 10.1097/01.prs.0000131021.17800.be. PMID 15318058
- [Background] Hatef DA, Brown SA, Lipschitz AH, Kenkel JM. Efficacy of lidocaine for pain control in subcutaneous infiltration during liposuction. Aesthet Surg J. 2009 Mar-Apr;29(2):122-8. doi: 10.1016/j.asj.2009.01.014. PMID 19371843
- [Background] Appelbaum N, Clarke J. Ideal body weight calculations: fit for purpose in modern anaesthesia? Eur J Anaesthesiol. 2021 Dec 1;38(12):1211-1214. doi: 10.1097/EJA.0000000000001515. No abstract available. PMID 33876785
- [Result] Mendez BM, Coleman JE, Kenkel JM. Optimizing Patient Outcomes and Safety With Liposuction. Aesthet Surg J. 2019 Jan 1;39(1):66-82. doi: 10.1093/asj/sjy151. PMID 29947738